CLINICAL TRIAL: NCT01850459
Title: Extracellular Signal-Related Kinase Biomarker Development in Autism
Acronym: ERK
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: CIN001- ERK in Autism
Record Dates: First submitted 2013-05-07; First posted 2013-05-09 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For the ERK activation assay, about 5 mL of whole blood is layered onto 3 mL Histopaque in a 15 mL centrifuge tube, and centrifuged. The lymphocyte-containing cell layer is removed and transferred for washing. After a second wash, cells are resuspended and rested. They are then stimulated by addition of phorbol myristate acetate and sample aliquots are removed at short intervals, fixed and permeabilized. Fixed, permeabilized cells are stained by addition of Alexafluor488-labeled monoclonal antibody to phospho-ERK in the dark for 30 min. Washed, resuspended cells are analyzed in a Coulter flow cytometer.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Autism Spectrum Disorder group: Diagnosis of autistic disorder as confirmed by a clinical interview, utilizing the DSM-V
- IQ-Matched Control Subjects
- Age-Matched Neurotypical Controls
- Shipped Biomarker Control Group Subjects: These subjects provide a blood sample only that serves as a shipping control that is shipped along with all blood samples from Autistic Disorder Subjects, IQ-Matched Control Subjects or Age-Matched Neurotypical Control Subjects. For these shipping control samples, blood samples will also be drawn from the subjects.

SUMMARY:
The purpose of this research study is to establish a way to help the development of targeted treatments in autism spectrum disorders. This may also help in early diagnosis of autism and may possibly predict severity. The study will compare subject's ERK (extracellular signal-related kinase) signaling to age- and gender-matched neurotypical controls and Intelligence quotient (IQ)-matched developmental disabilities.

DETAILED DESCRIPTION:
Autism Spectrum Disorder Subject Criteria:

Inclusion Criteria:

* Diagnosis of autism spectrum disorder, based upon a clinical interview utilizing the Diagnostic and Statistical Manual-V (DSM-V)
* Age 3-25 years
* Stable dosing of psychotropic drugs for greater than or equal to 5 half-lives

Exclusion Criteria:

* Diagnosis of schizophrenia, another psychotic disorder, bipolar disorder, or alcohol or other substance abuse based on Diagnostic and Statistical Manual-V criteria
* Use of lithium, riluzole or other known modulators of ERK activation

Age-Matched Neurotypical Control Subjects:

* Age matched to the age of an Autistic Disorder Subject
* History of normal development

IQ-Matched Control Subjects:

* Those subjects who are included in the study based on having an IQ and age that matches the IQ and age of an Autistic Disorder Subject who has an IQ less than 70
* All IQ-Matched Control Subjects will then also have an IQ less than 70

ELIGIBILITY:
Inclusion Criteria (ASD subjects):

* Diagnosis of autistic disorder as confirmed by a clinical interview, utilizing the DSM-V
* Age 3-25 years
* Stable dosing of psychotropic drugs for 5 half-lives or greater

Exclusion Criteria (ASD subjects):

* Diagnosis of schizophrenia, another psychotic disorder, bipolar disorder, or alcohol or other substance abuse based on DSM-V criteria
* Use of lithium, riluzole or other known modulators of ERK activation

IQ-Matched Control Subjects: Those subjects who are included in the study based on having an IQ and age that matches the IQ and age of an Autistic Disorder Subject who has an IQ less than 70. All IQ-Matched Control Subjects will then also have an IQ less than 70. IQ-Matched Control Subjects participate in a Screen/Baseline visit only.

Age-Matched Neurotypical Control Subjects: Those subjects who are included in the study based on having an age matched to the age of an Autistic Disorder Subject and a history of normal development. Age-Matched Neurotypical Subjects participate in a Screen/Baseline visit only.

Shipped Biomarker Control Group Subjects: For these shipping control samples, blood samples will also be drawn from adult parent/guardians of participating subjects.

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The subjects with autism will be recruited through the clinic population at Cincinnati Children's Hospital Medical Center. Recruitment of subjects will be conducted by notifying via, IRB approved electronic and paper ads, individuals with autistic disorder, their families, treating clinicians and agencies throughout the referral base of CCHMC and those within our existing clinical services, residential facilities, schools and group homes for the developmentally disabled.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2013-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
ERK activation | Up to three years

CONTACTS AND LOCATIONS:
Overall Officials: Craig A. Erickson, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States